CLINICAL TRIAL: NCT03073070
Title: Red Blood Cell Lifespan Measurement in Diabetic Children
Brief Title: RBC Lifespan Measurement in Diabetic Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guohua An (Other)
Responsible Party: Sponsor-Investigator, Guohua An, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201612763
Record Dates: First submitted 2016-12-18; First posted 2017-03-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Diabetes; Red Blood Cell Survival
Keywords: diabetic children; RBC lifespan
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biotin labeled RBCs in 4-10 year old diabetes children (Experimental): Biotin labeled autologous RBCs will be transfused to the subjects
  Interventions: Drug: biotin labeled RBCs
- Biotin labeled RBCs in 10-18 year old diabetes children (Experimental): Biotin labeled autologous red blood cells will be transfused to the subjects
  Interventions: Drug: biotin labeled RBCs

INTERVENTIONS:
Drug: biotin labeled RBCs — Autologous red blood cells are biotin labeled and transfused to the subjects. Survival of these red blood cells is tracked through examination of blood samples until no biotin-labeled red blood cells is detectable.
  Other Names: biotinylated RBCs

SUMMARY:
HbA1c, a measure of mean blood glucose over the lifespan of a red blood cell (RBC), is a marker of increasing importance both for assessing glycemic control in children with known diabetes and for the diagnosis of diabetes in children. HbA1c has demonstrated poor reliability in diagnosis and management of pediatric diabetes and the most plausible reason for this unreliability is that the reference ranges of HbA1c were established based on 120-day RBC lifespan observed in adults, without considering the RBC lifespan difference between children and adults. The proposed studies will for the first time determine RBC lifespan in diabetic children

DETAILED DESCRIPTION:
Screening visit: There will be one screening visit before the study. We will do some blood tests that will determine if the subjects can be in this study. If the subject is qualify, he/she will be asked to return for the following scheduled visits.

Study visit 1: We will draw a small amount of subject's blood from the IV. The study subject's blood will then be marked with biotin. We will give back the subject's blood marked with biotin through IV within 4 to 6 hours. Endotoxin analysis (conducted pre-infusion) and bacterial culture analysis (conducted post-infusion) will be performed. Twenty minutes after the blood transfusion, we will draw blood from the IV. After that, we will take out the IV and the subject can go home.

All follow-up study visits:

The subject will have a study visit 24 hours after receiving blood marked with biotin. After that, the subject will have a clinic visit every 7-10 days. These visits will end when we can no longer find the biotin marked blood cells in the subject's blood. This is expected to be approximately 12 weeks later.

At these visits, we will draw blood and also collect all blood glucose results in the past 7-10 days.

After the study visits are completed, there will be one follow-up visit 4-6 months after the subject receives the biotin marked RBCs. We will draw about 0.25 ml of blood.

Continuous glucose monitoring and HbA1c determination-- We will monitor continuous glucose concentrations throughout the study. This will be accomplished by setting up FreeStyle Libre Pro continuous glucose monitoring (CGM) device for each study subject. In addition, HbA1c will be measured once in the middle of the study (likely visit 6) and in the end of the study (likely visit 12).

ELIGIBILITY:
Inclusion Criteria:

* children with either type1 or type 2 diabetes between 4-18 years old

Exclusion Criteria:

* consumption of biotin supplements or raw eggs within 30 days;
* history of gastrointestinal blood loss;
* heart failure ;
* active viral or bacterial infection;
* hemoglobinopathy;
* prior history of liver disease with transaminases more than 3 times the upper limit of normal for age;
* uncontrolled thyroid disease;
* anemia (whole blood HCT<33);
* history of renal disease (prior serum creatinine more than >1.5 mg/dlL);
* detectable antibody to biotin.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Measurement of RBC survival in diabetic children using biotin-labeled RBCs | 50 days to 120 days
  the lifespan of red blood cells in children with diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Guohua An, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No